CLINICAL TRIAL: NCT06316323
Title: The Effect of Silver Diamine Fluoride and Sodium Fluoride Varnish on Salivary pH and Streptococcus Mutans and Lactobacillus in Early Childhood Caries: A Randomized Control Trial
Brief Title: The Anticariogenic Effect of Silver Diamine Fluoride and Sodium Fluoride Varnish
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Nur Amalina Asmad, Dr, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/09/2021 (FB/51)
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Early Childhood Caries
Keywords: silver diamine fluoride; fluoride varnish; early childhood caries
MeSH Terms: interventions — silver diamine fluoride; Sodium Fluoride

STUDY DESIGN:
Intervention Model Description: one group received silver diamine fluoride treatment, and another group received sodium fluoride varnish treatment
Who Masked: Outcomes Assessor
Masking Description: Subjects that participated in this study were randomly allocated to two groups; Group A and Group B. Group A subjects were treated with 38% SDF and Group B subjects were treated with 5% NaF varnish. The randomisations of the subjects were done using a sealed envelope. Sequentially numbered, opaque sealed envelopes (SNOSE) method was used for the allocation concealments. This study was conducted in a non-blinded manner, as it was deemed impossible to blind the subjects. The treatment solutions utilized in this study were clearly distinct, with the SDF solution comprising a two-step process, while NaF varnish only required a single step. Additionally, the treatments exhibited different colors and textures. Consequently, the principal investigator had to closely supervise the treatment of each group. Due to the risk of blackish staining associated with SDF, parents and children were not blinded and were informed of the treatment they would receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Silver Diamine Fluoride
  Interventions: Drug: Silver diamine fluoride
- Group B (Experimental): Sodium Fluoride Varnish
  Interventions: Drug: Sodium fluoride

INTERVENTIONS:
Drug: Silver diamine fluoride — 38% Silver Diamine Fluoride (SDF) is a topical antimicrobial and remineralizing agent which was cleared by the FDA as a Class II medical device to treat tooth sensitivity. In certain circumstances, SDF may be used as a non-restorative treatment to arrest carious lesions on primary and permanent teeth
  Other Names: SDF
  Arms: Group A
Drug: Sodium fluoride — Fluoride varnish to apply on tooth surface, so that the tooth becomes more resistant to caries attack. The active ingredient of fluoride varnish is 5% sodium fluoride, (22,600 ppm fluoride)
  Other Names: NaF
  Arms: Group B

SUMMARY:
Sodium Fluoride (NAF) varnish was considered as the treatment of Early Childhood Caries (ECC). However, the emergence of Silver Diamine Fluoride (SDF) has become more popular to tackle dental caries among children. SDF has silver ions that harbor antibacterial properties that play a crucial role in arresting active, cavitated carious lesions and has fluoride ions that are important in remineralizing enamel and dentin. This randomized control trial aims to compare the effect of SDF and NaF varnish on the salivary pH and density of Streptococcus mutans and Lactobacillus. 49 subjects below 6 years old, attending dental treatment at the Faculty of Dentistry, Universiti Teknologi MARA (UiTM) were recruited and were divided into two groups of treatment: 38% SDF or 5% SDF. Saliva samples of each subject were collected to test for salivary pH and density of S. mutans and Lactobacillus before the treatment and after 3 months of treatment. The salivary pH were tested using a calibrated pH meter. Saliva samples were subjected to microbiological analysis using Colony Forming Unit (CFU) and quantitative Polymerase Chain Reaction (qPCR) technique. The findings of this study will be used to support the use of SDF as an alternative to NaF varnish and to develop a recommendation guideline on the clinical use of SDF in ECC management.

DETAILED DESCRIPTION:
ECC continues to become a significant oral health concern owing to its high prevalence worldwide despite the preventive measures taken, including excessive oral health promotion. While conventional tooth restoration has been widely accepted as a standard intervention in managing ECC, the traumatic effects it causes may lead to dental fear, which prevents children from receiving dental treatment and subsequently leads to caries sequelae and complications. There is well-established evidence-based research proving the benefits of fluoride-based products in preventing dental caries. Previously, caries prevention in ECC was widely considered to be due to sodium fluoride (NaF) varnish. However, a systematic review found that treating dental caries with 5% NaF varnish is insufficient, urging the need to find another solution that is effective in halting caries progression.

In recent years, there has been great interest in the use of Silver Diamine Fluoride (SDF) as a new method for caries prevention because of its superior effects. The utilisation of SDF eliminates the necessity for tooth drilling, and it possesses anticariogenic properties that are essential for curbing active and cavitated carious lesions by rebuilding enamel and dentin. Existing data indicate that employing a non-invasive method of applying SDF with a 38% concentration twice a year can effectively manage ECC by up to 76.3% after a 30-month follow-up period. The application of 38% SDF has been demonstrated to significantly reduce the occurrence of new caries in treated children by approximately 77% compared with non-treated children.

Although various mechanisms underlying the antibacterial effects of SDF have been elucidated, data on its effects on salivary pH and cariogenic bacteria, particularly S. mutans and Lactobacillus, are lacking. Although several in vivo studies have explored the effect of SDF on S. mutans and Lactobacillus, the scarcity of clinical investigations remains a challenge. This study provides a better understanding of the effects of SDF on the modulation of salivary pH and S. mutans and Lactobacillus and provides scientific evidence on the mechanism of action of SDF in the oral environment. Therefore, this study is crucial to support the use of SDF in clinical settings as an alternative to the conventional method of treatment in managing ECC. To date, there is no clinical data regarding the use of SDF in Malaysia or the investigation of cariogenic bacterial profiling following SDF treatment among the Malaysian population. therefore the general research objective is to compare the effects of 38% SDF and 5% NaF on salivary pH, S. mutans, and Lactobacillus counts in children with ECC.

ELIGIBILITY:
Inclusion Criteria:

* Children under 6 years old, with ECC, having at least one active dentinal caries were included in this study. The cavitated tooth was assessed using International Caries Detection and Assessment System (ICDAS). Children that only had the tooth that fulfilled the ICDAS score 5 were included. This is characterized by a distinct cavity with visible dentine, not including more than half of the tooth. The tooth must not be mobile, associated with abscess, or have the symptoms of irreversible pulpitis. Children that had been included in this study must have not been on antibiotic treatment for at least 3 months before the start of the study and not being put on such treatment throughout the study period

Exclusion Criteria:

* Children with any severe medical conditions, emotional or physical disorders were excluded from the study. Children that had been using chlorhexidine mouthwashes within 2 weeks before the baseline appointment or professional topical fluoride was applied in the past 6 months were also excluded. Another exclusion criteria are children that had gingival or perioral ulceration or stomatitis, or a tooth abscess, have a history of chemical allergies to silver, fluoride, potassium, iodine, and ammonia, and uncooperative child. Besides that, parents and children that were refused any type of treatment were excluded. Children who did not complete the follow up were considered dropouts.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-01-26 (Actual)

PRIMARY OUTCOMES:
comparison of salivary pH | 3 months
  to compare the salivary pH before and after 3 months of 38% SDF and 5% NaF treatment
comparison of salivary counts of Streptococcus mutans | 3 months
  to compare the salivary counts of Streptococcus mutans before and after 3 months of 38% SDF and 5% NaF treatment
comparison of salivary counts of Lactobacillus | 3 months
  to compare the salivary counts of Lactobacillus before and after 3 months of 38% SDF and 5% NaF treatment

SECONDARY OUTCOMES:
Detection and comparison of salivary counts of Lactobacillus acidophilus | 3 months
  to compare the relative numbers of Lactobacillus acidophilus before and after 3 months of 38% SDF and 5% NaF treatment with qPCR

CONTACTS AND LOCATIONS:
Overall Officials: NUR ASMAD, BDS, MScD, Principal Investigator — University Technology MARA
Locations (1):
- University Technology MARA, Sungai Buloh, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No